CLINICAL TRIAL: NCT01746862
Title: A Randomized, Open-label, Two-arm Parallel Group, No Treatment Group-controlled, Multicenter Phase III Study to Evaluate the Safety and Efficacy of Saizen® 0.067 mg/kg/Day Subcutaneous Injection in Children With Idiopathic Short Stature
Brief Title: A Phase 3 Study to Evaluate the Safety and Efficacy of Saizen® in Children With Idiopathic Short Stature (ISS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200104-533
Record Dates: First submitted 2012-11-30; First posted 2012-12-11 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-08

CONDITIONS: Idiopathic Short Stature
Keywords: Saizen®; Recombinant human growth hormone (r-hGH); Idiopathic short stature; Height velocity; Bone age
MeSH Terms: interventions — Human Growth Hormone

ARMS (2):
- Saizen Test Group (Experimental)
  Interventions: Drug: Saizen®
- Saizen Control Group (Active Comparator)
  Interventions: Drug: Saizen®

INTERVENTIONS:
Drug: Saizen® — Subjects in the Saizen test group will receive Saizen (recombinant-human growth hormone [r-hGH]) subcutaneously 6 days per week at a weight based dose of 0.067 milligram per kilogram of body weight per day (mg/kg/day) for 12 months.
  Other Names: Somatropin; r-hGH
  Arms: Saizen Test Group
Drug: Saizen® — Subjects in the Saizen control group will receive no treatment for the first 6 months and thereafter will receive Saizen (r-hGH) subcutaneously 6 days per week at a weight based dose of 0.067 mg/kg/day for the next 6 months.
  Other Names: Somatropin; r-hGH
  Arms: Saizen Control Group

SUMMARY:
This is an open-label, multi-center, randomized, two-arm parallel, no-treatment group controlled (only for the first 6 months), Phase 3 study in children with ISS. The subjects will be treated with 0.067 milligram/kilogram/day (mg/kg/day) of Saizen®, weight base dose, for 12 months (12 months of treatment in the test group, and 6 months of no treatment and then 6 months of treatment in the control group).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 5 years
* Pre-pubertal; testicular volume less than 4 milliliter (in males) and breast Stage 1 (in females)
* The official records of height (for example records measured in hospitals or schools) during previous 6 months or more preceding inclusion in the study (self-measurement of the height at home will not be considered as a valid record)
* Height less than or equal to 3rd percentile compared to same sex, same age
* Peak serum growth hormone (GH) greater than 10 microgram per liter (mcg/L) in GH stimulation test (results of peak serum GH greater than 10 mcg/L in GH stimulation test within 1 year can be used instead)
* Naive to GH therapy
* Normal birth weight (that is greater than or equal to 3rd percentile when compared to same sex)
* Normal thyroid function
* Normal karyotype in girls
* Written informed consent from parent/guardian
* Written informed consent from the subject who speaks, understand, read, and write Korean
* Bone age less than 10 years in boys and less than 9 years in girls, whose difference between the bone and chronological age is no more than 3 years

Exclusion Criteria:

* Puberty development (Tanner stage greater than or equal to 2)
* Skeletal dysplasia or abnormal body proportions
* Chronic systemic illness
* Dysmorphic syndrome
* Growth Hormone Deficiency
* Small for Gestational Age (SGA)
* Current medication for Attention deficit hyperactivity disorder (ADHD) or hyperactivity disorder
* Current medication with drugs that may influence secretion or action of growth hormone (such as estrogen, androgen, anabolic steroid, corticosteroid, thyroxine, aromatase inhibitors)
* Diabetes mellitus
* Kidney transplantation
* Acute critical illness, including complications following open heart surgery, abdominal surgery or multiple accidental trauma
* Acute respiratory failure
* Malignancy or previous therapy for malignancy
* Known hypersensitivity to somatotropin or any of its excipients including cresol or glycerol
* Closed epiphyses, progression or recurrence of an underlying intracranial tumor, chronic renal disease
* Endocrinologic or metabolic disorders such as Prader-Willi syndrome; Russel-Silver syndrome; Seckel syndrome; Down syndrome; Cushing syndrome; Noonan syndrome; short stature caused by other chromosomal abnormalities
* The disorders that explain short stature such as psychiatric disorders, nutritional disorders, and chronic debilitating diseases
* Participation in another clinical trial within the past 3 months
* Status of legal incapacity or limited legal capacity of the parents or legal guardian

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Ltd.
Locations (1):
- Please contact Merck KGaA Communication Center for Recruiting Sites, Located in, South Korea

REFERENCES:
- [Derived] Chung WY, Yoo HW, Hwang JS, Ko CW, Kim HS, Jin DK, Lee KH, Han HS, Paranchothy P, Suh BK. Effect of Growth Hormone Therapy on Height Velocity in Korean Children with Idiopathic Short Stature: A Phase III Randomised Controlled Trial. Horm Res Paediatr. 2018;90(1):44-53. doi: 10.1159/000491016. Epub 2018 Aug 15. PMID 30110706

RESULTS

PARTICIPANT FLOW:
Groups:
- Saizen Test Group: Subjects in the Saizen test group received Saizen (recombinant-human growth hormone [r-hGH]) subcutaneously 6 days per week at a weight based dose of 0.067 milligram per kilogram of body weight per day (mg/kg/day) for 12 months.
- Saizen Control Group: Subjects in the Saizen control group received no treatment for the first 6 months and thereafter received Saizen (r-hGH) subcutaneously 6 days per week at a weight based dose of 0.067 mg/kg/day for the next 6 months.
Period: Overall Study
Arm/Group | Saizen Test Group | Saizen Control Group
Started | 60 | 30
Treated | 59 | 30
Completed | 52 | 27
Not Completed | 8 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Consent withdrawal by parent's guardian | 5 | 2
Not completed — Entered puberty during the study | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) included all randomized subjects who received at least 1 dose of planned trial treatment and had follow-up safety data. SAS also included the safety data for all subjects during non-treatment (the first 6 months after enrollment) period who belonged to control group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Saizen Test Group | Saizen Control Group | Total
Number analyzed (Participants) | 59 | 30 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.79 (1.54) | 6.83 (1.61) | 6.80 (1.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 13 | 42
  Male | 30 | 17 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Height Velocity at Month 6 Using Last Observation Carried Forward (LOCF) Method
Description: Baseline height is defined as the last available height measurement before randomization. Baseline height velocity = ([Baseline height minus height measurement obtained at least 6 months prior] / 6) * 12. Height velocity at Month 6 = ([Month 6 height minus height measurement obtained at least 6 months prior] / 6) * 12.
Time Frame: Baseline, Month 6
Population: Intent-to-treat (ITT) analysis set included all randomized subjects, regardless of whether or not they received the treatment to which they were randomized, completed the study or had any protocol deviations. Here "n" signifies those subjects who were evaluable for this outcome measure at the specified time points.
Measure: Mean (Standard Deviation); unit: centimeter/year (cm/yr)
Arm/Group | Saizen Test Group | Saizen Control Group
Number analyzed (Participants) | 60 | 30
centimeter/year (cm/yr)
  Baseline (n=59,30) | 5.63 (1.62) | 4.94 (1.91)
  Change at Month 6 (n=59,29) | 4.45 (2.70) | 1.01 (3.15)
Statistical Analysis 1: Comparison: Saizen Test Group vs Saizen Control Group; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis was performed using analysis of covariance (ANCOVA) with baseline age and baseline height as the covariates; Least Squares (LS) Mean Difference = 3.47, 95% CI 2-sided [2.17 to 4.78]

2. Secondary Outcome: Change From Baseline in Height Velocity at Month 12
Description: Baseline height is defined as the last available height measurement before randomization. Baseline height velocity = ([Baseline height minus height measurement obtained at least 12 months prior] / 12) * 12. Height velocity at Month 12 = ([Month 12 height minus height measurement obtained at least 12 months prior] / 12) * 12.
Time Frame: Baseline, Month 12
Population: ITT analysis set included all randomized subjects, regardless of whether or not they received the treatment to which they were randomized, completed the study or had any protocol deviations. Here "Number of participants analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Saizen Test Group | Saizen Control Group
Number analyzed (Participants) | 52 | 27
cm/year | 3.77 (2.21) | 2.86 (1.95)

3. Secondary Outcome: Change From Baseline in Height at Month 6 and 12
Time Frame: Baseline, Month 6, Month 12
Population: ITT analysis set included all randomized subjects, regardless of whether or not they received the treatment to which they were randomized, completed the study or had any protocol deviations. Here "n" signifies those subjects who were evaluable for this outcome measure at the specified time points.
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Saizen Test Group | Saizen Control Group
Number analyzed (Participants) | 60 | 30
centimeter (cm)
  Baseline (n=60, 30) | 108.27 (7.67) | 108.07 (8.36)
  Change at Month 6 (n=55, 27) | 5.41 (1.04) | 3.10 (0.84)
  Change at Month 12 (n=52, 27) | 9.78 (1.35) | 8.24 (1.47)

4. Secondary Outcome: Change From Baseline in Height Standard Deviation Score (SDS) at Month 6 and 12
Description: Height SDS was calculated as: Height SDS = (measured height - population mean) / population standard deviation, where mean and standard deviation were based on the Korean standard growth charts. SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) a subject's value was relative to the mean of the reference population. The scores were centred around zero. Negative score indicated a subject was smaller for their age/gender.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Saizen Test Group | Saizen Control Group
Number analyzed (Participants) | 60 | 30
standard deviation score
  Baseline (n=60,30) | -2.26 (0.36) | -2.34 (0.34)
  Change at Month 6 (n=55, 27) | 0.59 (0.21) | 0.08 (0.19)
  Change at Month 12 (n=52, 27) | 0.96 (0.27) | 0.62 (0.27)

5. Secondary Outcome: Change From Baseline in Serum Concentration of Insulin-like Growth Factor-I (IGF-I) at Month 6 and 12
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microgram/liter (mcg/L)
Arm/Group | Saizen Test Group | Saizen Control Group
Number analyzed (Participants) | 60 | 30
microgram/liter (mcg/L)
  Baseline (n=60,30) | 112.62 (43.06) | 125.01 (65.68)
  Change at Month 6 (n=55, 27) | 122.57 (96.99) | 8.30 (41.57)
  Change at Month 12 (n=52, 27) | 164.48 (95.69) | 142.17 (112.94)

6. Secondary Outcome: Change From Baseline in Serum Concentration of Insulin Like Growth Factor Binding Protein-3 (IGFBP-3) at Month 6 and 12
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Saizen Test Group | Saizen Control Group
Number analyzed (Participants) | 60 | 30
mcg/L
  Baseline (n=60, 30) | 3,783.33 (915.20) | 3,935.67 (866.42)
  Change at Month 6 (n=55, 27) | 857.64 (761.28) | -38.89 (616.88)
  Change at Month 12 (n=52, 27) | 932.31 (666.13) | 545.56 (599.52)

7. Secondary Outcome: Percentage of Adherence to Study Treatment
Description: Percentage of adherence to study treatment (adherence rate) was defined as the actual number of received treatments divided by the scheduled number of treatments multiplied by 100. The adherence rate for 6 months was calculated from Baseline to 6 months for the Saizen Test Group and from Month 6 to Month 12 for the Saizen Control Group.
Time Frame: 6 months post-dose (Saizen Test Group and Saizen Control Group); 12 months post-dose (Saizen Test Group)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of adherance
Arm/Group | Saizen Test Group | Saizen Control Group
Number analyzed (Participants) | 60 | 30
percentage of adherance
  Adherence for 6 months (n=60, 27) | 94.38 (14.12) | 95.69 (5.04)
  Adherence for 12 months (n=60, 0) | 93.27 (14.67) | NA (NA) — Data was not available as control group received the treatment for only 6 months

8. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence which does not necessarily have a causal relationship with this the study drug. An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. For the Saizen Test Group, TEAEs were defined as events that occurred or worsened at or after the first administration of treatment and for the Saizen Control Group, TEAEs were defined as events that occurred or worsened at or after the randomization.
Time Frame: Baseline up to Month 13
Population: as for baseline characteristics
Measure: Number; unit: subjects
Groups:
- Saizen Test Group; Saizen Control Group: Subjects in the Saizen control group received no treatment for the first 6 months and thereafter received Saizen (r-hGH) subcutaneously 6 days per week at a weight based dose of 0.067 mg/kg/day for the next 6 months.
Arm/Group | Saizen Test Group | Saizen Control Group
Number analyzed (Participants) | 59 | 30
subjects
  TEAEs | 42 | 18
  Serious TEAEs | 3 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Month 13
Description: Safety analysis set (SAS) included all randomized subjects who received at least 1 dose of planned trial treatment and had follow-up safety data. SAS also included the safety data for all subjects during non-treatment (the first 6 months after enrollment) period who belonged to control group.
Arm/Group | Saizen Test Group | Saizen Control Group
Serious Adverse Events (participants affected / at risk) | 3/59 | 1/30
Other Adverse Events (participants affected / at risk) | 42/59 | 18/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saizen Test Group (N=59) | Saizen Control Group (N=30)
Pyrexia (General disorders) | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Chronic tonsillitis (Infections and infestations) | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saizen Test Group (N=59) | Saizen Control Group (N=30)
Motion sickness (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Pectus carinatum (Congenital, familial and genetic disorders) | 1 | 0
Chalazion (Eye disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1
Eye inflammation (Eye disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Oral mucosal eruption (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 24 | 9
Upper respiratory tract infection (Infections and infestations) | 14 | 9
Rhinitis (Infections and infestations) | 4 | 2
Bronchitis (Infections and infestations) | 2 | 3
Conjunctivitis (Infections and infestations) | 4 | 0
Gastroenteritis (Infections and infestations) | 4 | 0
Otitis media (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 2 | 1
Acute tonsillitis (Infections and infestations) | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Molluscum contagiosum (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0
Perineal infection (Infections and infestations) | 1 | 0
Pulpitis dental (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tinea infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No